CLINICAL TRIAL: NCT01373736
Title: 123I-MIBG Scintigraphy in Patients Being Evaluated for Neuroendocrine Tumors
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vancouver Coastal Health (Other Government)
Responsible Party: Daniel Worsley, Vancouver Coastal Health
Purpose: Diagnostic
Other Study IDs: H10-02695
Record Dates: First submitted 2011-06-13; First posted 2011-06-15 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Pheochromocytoma; Neuroblastoma; Paraganglioma; Medullary Thyroid Carcinoma; Carcinoid Tumors
MeSH Terms: conditions — Pheochromocytoma; Neuroblastoma; Paraganglioma; Carcinoma, Medullary; Carcinoid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: 123I-meta-iodobenzylguanidine

SUMMARY:
The study is designed to study the safety and effectiveness of 123I-MIBG as a diagnostic imaging agent in evaluating patients with known or suspected neuroendocrine tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a clinical indication for 123I-MIBG imaging to evaluate for the presence, extent, or status of neuroendocrine tumors;
* subjects must be able and willing to comply with study procedures.

Exclusion Criteria:

* Subjects with history of renal insufficiency (serum creatinine level > 3.0 mg/dL [265 µmol/L]) and inability to be withdrawn from medications known to interfere with 123I-MIBG uptake;
* Subjects unable to tolerate lying supine;
* Subjects pregnant or breastfeeding, unless the information to be gained outweighs the possible hazardous effects of 123I-MIBG administration. Where the assessment of the risk/benefit ration suggests the use of 123I-MIBG in nursing mothers, the breastfeeding should be discontinued for at least 48 hours post-injection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Worsley, MD, Principal Investigator — Vancouver Coastal Health
Locations (1):
- Vancouver Coastal Health, Vancouver, British Columbia, Canada